CLINICAL TRIAL: NCT04887285
Title: Can Distraction Substitute for Procedural Sedation and Improve Tolerance in Patients Receiving Epidural Steroid Injection for Pain? A Randomized Controlled Trial
Brief Title: Virtual Reality as a Substitute for Procedural Sedation During Epidural Steroid Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Geneva Foundation (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00255275; HU00011920011 (Other Grant/Funding Number: Department Of Defense)
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Lower Back Pain; Lumbar Radiculopathy
Keywords: epidural steroid injection; virtual reality; distraction; sedation; lumbar radiculopathy
MeSH Terms: conditions — Low Back Pain; Radiculopathy | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel study comparing virtual reality to sedation to standard care (no sedation or virtual reality) for procedure-related pain in patients undergoing lumbar epidural steroid injections.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be unaware of treatment allocation but the patient and provider cannot be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Virtual reality (VR) (Experimental): Subjects in the VR group will be fitted with an HTC headset and headphones with disposable ear covers. They will choose from a menu of 6 different programs. They will also receive 1% superficial anesthesia.
  Interventions: Device: Virtual reality
- Sedation (Active Comparator): Conscious sedation will be accomplished by the use of midazolam and/ or fentanyl. We will use a wide range of dosing (1-5 mg for midazolam, up to 150 mcg for fentanyl) to maximize generalizability and account for widespread variability in clinical circumstances, medical practice and patient response (personalized medicine). All medications will be titrated to conscious sedation by a board-certified anesthesiologist. Subjects will also receive 1% superficial anesthesia.
  Interventions: Drug: Intravenous sedation
- Standard care (Other): Patients in this arm will be administered only 1% lidocaine as superficial anesthesia, similar to the other 2 arms.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Virtual reality — Subjects in the virtual reality group will be offered a variety of immersive environments to choose from (mountains, beach, rainforest and temperate forest) in addition to local anesthetic.
  Arms: Virtual reality (VR)
Drug: Intravenous sedation — Sedation will be administered using low-dose midazolam and/ or fentanyl. We will use a wide range of dosing (1-5 mg for midazolam, up to 150 mcg for fentanyl) to maximize generalizability and account for widespread variability in clinical circumstances, medical practice and patient response (personalized medicine). Sedation will be titrated to effect by a board-certified or eligible anesthesiologist so that patients remain responsive to verbal stimuli.
  Arms: Sedation
Other: Standard care — Patients will receive superficial local anesthetic with 1% lidocaine. Local anesthetic will be administered by the physician performing the procedure titrated to patient comfort.
  Other Names: Local anesthetic only
  Arms: Standard care

SUMMARY:
This study examines the impact of virtual reality compared to sedation (midazolam and/or fentanyl) and no intervention on pain experienced from an epidural steroid injection (ESI). The intervention group (who receive virtual reality as a distraction modality) is compared to a sedation group and a control group.

DETAILED DESCRIPTION:
All patients enrolled in the study will already be undergoing lumbar epidural steroid injections for lumbar radicular pain as part of their clinical care. The epidural approach will either be transforaminal or interlaminar depending on clinical judgment (i.e. transforaminal ESI for unilateral pain, interlaminar ESI for bilateral pain). The study will consist of 3 groups: virtual reality, sedation, and a control group which receives no intervention (i.e. standard of care). The virtual reality group will receive virtual reality via a headset containing a menu of 6 programs that the subject can choose; the sedation group will receive from 1-5 mg of midazolam and up to 150 mcg of fentanyl as clinically indicated, and the control group will not receive an intervention (standard of care). All subjects will also receive 1% lidocaine local anesthetic through a 25-gauge needle for superficial anesthesia, which is standard of care. Subjects will be randomized to each of these groups, with sub-allocation being done stratified by the type of ESI (transforaminal vs. interlaminar).

A secondary pilot study will evaluate whether a processed electroencephalogram (pEEG) and continuous colored density spectral array monitored via a four-channel Masimo SEDLine frontal EEG sensor can serve as a biomarker for painful stimulation and the effectiveness of distraction and sedation to reduce acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and females; ages 18-90 years
* Lumbosacral radicular pain with a baseline average of leg pain score of > 4/10, MRI findings (if available) consistent with symptoms, duration of pain > 6 weeks, and no previous lumbar spine surgery.
* Documented diagnosis of radicular pain caused by herniated disc, central stenosis, foraminal stenosis, degenerative disk disease
* Willingness to adhere to undergo ESI with either sedation (midazolam and or fentanyl) or with virtual reality
* Able to appear for a follow up visit between 24-40 days following the intervention

Exclusion Criteria:

* MRI findings discordant with symptoms (absence of herniated disc, spinal stenosis or severe disc degeneration without nerve root impingement (e.g. annular tears) that could explain symptoms)
* Previous lumbosacral spine surgery at the area affected
* Prior ESI within the past 6 months
* Allergy to contrast dye
* Poorly controlled psychiatric conditions that could affect outcomes (e.g. active substance abuse) or impose a barrier to participation (e.g. anxiety disorder requiring procedural sedation)
* Morbid obesity (BMI >40)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Whitley Lucio, Study Director — Walter Reed National Military Medical Center; Steven P Cohen, MD, Principal Investigator — Johns Hopkins Uinversity - SOM Ane Pain; Nuj Tontisirin, MD, Study Director — Ramathibodi Hospital, Mahidol University; Pornpan Chalermkitpanit, MD, Study Director — King Chulalongkorn Memorial Hospital, Chulalongkorn University; Pramote Euasobhon, MD, Study Director — Siriraj Hospital; Sithapan Munjupong, MD, Study Director — Phramongkutklao College of Medicine; Qian Chen, MD, Study Director — NYU Langone Health
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol, Informed Consent Form, deidentified data and statistical code.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication until 3 years
Access Criteria: By e-mail request, upon approval by Dept. of Defense

REFERENCES:
- [Result] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Result] Mallari B, Spaeth EK, Goh H, Boyd BS. Virtual reality as an analgesic for acute and chronic pain in adults: a systematic review and meta-analysis. J Pain Res. 2019 Jul 3;12:2053-2085. doi: 10.2147/JPR.S200498. eCollection 2019. PMID 31308733

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality (VR): Subjects in the VR group will be fitted with an HTC headset and headphones with disposable ear covers. They will choose from a menu of 6 different programs. The participants will also receive 1% superficial anesthesia.
  Virtual reality: Subjects in the virtual reality group will be offered a variety of immersive environments to choose from (mountains, beach, rainforest and temperate forest) in addition to local anesthetic.
- Sedation: Conscious sedation will be accomplished by the use of midazolam and/ or fentanyl. The investigators will use a wide range of dosing (1-5 mg for midazolam, up to 150 mcg for fentanyl) to maximize generalizability and account for widespread variability in clinical circumstances, medical practice and patient response (personalized medicine). All medications will be titrated to conscious sedation by a board-certified anesthesiologist. Subjects will also receive 1% superficial anesthesia.
  Intravenous sedation: Sedation will be administered using low-dose midazolam and/ or fentanyl. The investigators will use a wide range of dosing (1-5 mg for midazolam, up to 150 mcg for fentanyl) to maximize generalizability and account for widespread variability in clinical circumstances, medical practice and patient response (personalized medicine). Sedation will be titrated to effect by a board-certified or eligible anesthesiologist so that patients remain responsive to verbal stimuli.
Period: Overall Study
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Started | 48 | 50 | 48
Completed | 48 | 48 | 45
Not Completed | 0 | 2 | 3
Not completed — Lost to Follow-up | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Virtual Reality (VR): Subjects in the VR group will be fitted with an HTC headset and headphones with disposable ear covers. The subjects will choose from a menu of 6 different programs. The subjects will also receive 1% superficial anesthesia.
  Virtual reality: Subjects in the virtual reality group will be offered a variety of immersive environments to choose from (mountains, beach, rainforest and temperate forest) in addition to local anesthetic.
- Total: Total of all reporting groups
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care | Total
Number analyzed (Participants) | 48 | 50 | 48 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 58 (13) | 56 (16) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 27 | 95
  Male | 17 | 13 | 21 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 47 | 50 | 47 | 144
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 26 | 22 | 25 | 73
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 17 | 13 | 39
  White | 12 | 7 | 8 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 31 | 29 | 87
  Thailand | 21 | 19 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Pain Score During Procedure
Description: 0-10 verbal rating scale (higher scores indicate greater pain)
Time Frame: Immediately after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Virtual Reality (VR): Subjects in the VR group will be fitted with an HTC headset and headphones with disposable ear covers. The subjects will choose from a menu of 6 different programs. They will also receive 1% superficial anesthesia.
  Virtual reality: Subjects in the virtual reality group will be offered a variety of immersive environments to choose from (mountains, beach, rainforest and temperate forest) in addition to local anesthetic.
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
score on a scale | 3.7 (2.5) | 3.2 (3.0) | 5.2 (3.1)

2. Secondary Outcome: Amount of Local Anesthetic Required
Description: Volume of 1% lidocaine used to complete the skin wheel prior to the procedure.
Time Frame: At the start of the procedure
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
milliliters | 5.6 (2.5) | 5.4 (2.6) | 6.3 (2.9)

3. Secondary Outcome: Subcutaneous Skin Wheal Pain Score
Description: 0-10 verbal rating scale (higher scores indicate greater pain)
Time Frame: Immediately after skin wheal
Population: Skin wheels were unintentionally omitted in two participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Virtual Reality (VR): Subjects in the VR group will be fitted with an HTC headset and headphones with disposable ear covers. Subjects will choose from a menu of 6 different programs. Subjects will also receive 1% superficial anesthesia.
  Virtual reality: Subjects in the virtual reality group will be offered a variety of immersive environments to choose from (mountains, beach, rainforest and temperate forest) in addition to local anesthetic.
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 49 | 47
score on a scale | 4.0 (2.4) | 3.8 (2.8) | 4.5 (2.8)

4. Secondary Outcome: Procedure Satisfaction
Description: This outcome was measured using a standalone question using the 1-5 Likert scale (1= very unsatisfied, 3= neither satisfied nor dissatisfied, 5= very satisfied). A mean of the participant selection is reported.
Time Frame: In postanesthetic care unit (within 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
score on a scale | 4.7 (0.6) | 4.6 (0.8) | 4.5 (0.7)

5. Secondary Outcome: Ability to Communicate
Description: This outcome was measured using a standalone question using the 1-5 Likert scale (1= complete inability to communicate, 2= markedly decreased ability to communicate, 3= slightly decreased ability to communicate, 4= no change in ability to communicate, 5= improved ability to communicate). A mean of the participant selection is reported.
Time Frame: In postanesthetic care unit (within 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Virtual Reality (VR): Subjects in the VR group will be fitted with an HTC headset and headphones with disposable ear covers. Subjects will choose from a menu of 6 different programs. The subjects will also receive 1% superficial anesthesia.
  Virtual reality: Subjects in the virtual reality group will be offered a variety of immersive environments to choose from (mountains, beach, rainforest and temperate forest) in addition to local anesthetic.
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
score on a scale | 4.1 (0.5) | 3.7 (0.9) | 4.0 (0.4)

6. Secondary Outcome: Procedure-related Anxiety
Description: This outcome was measured using a standalone question using the 1-5 Likert scale (1=extreme anxiety, 2=high anxiety, 3=average or expected anxiety, 4=minimal or mild anxiety, 5=no anxiety. A mean of the participant selection is reported.
Time Frame: In postanesthetic care unit (within 1 hour)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
score on a scale | 4.0 (1.3) | 4.2 (1.1) | 3.8 (1.1)

7. Secondary Outcome: Time to Discharge From Postanesthetic Care Unit
Description: Time to discharge from postanesthetic care unit, in minutes
Time Frame: At discharge from postanesthetic care unit assessed up to 6 hours
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
minutes | 27.0 [21.0 to 33.0] | 38.8 [34.7 to 42.9] | 24.4 [17.4 to 31.4]

8. Secondary Outcome: Participants With Positive Categorical Outcome
Description: This outcome measure is either positive or negative. A positive outcome is measured by participants with a 2-point or greater reduction in average leg pain score coupled with participants with a score of 5 or greater score on the Patient Global Impression of Change (PGIC), or negative is measure by a 1 or no point reduction in the average leg pain score couple with a 4 or less score on the Patient Global Impression of Change (PGIC). The average leg pain score on 0-10 numerical rating scale over the last week (higher pain scores indicate greater pain). The Patient global impression of change on 7-point Likert scale (from 1= no change, 3= a little better 5= moderately better, a slight but noticeable change, to 7=a great deal better, a considerable improvement that has made all the difference). Participants with positive outcome are reported.
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
Participants | 25 | 25 | 24

9. Secondary Outcome: Average Leg Pain Score
Description: Average leg pain score on 0-10 numerical rating scale over the last week (higher pain scores indicate greater pain)
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 3.0 (2.4) | 3.1 (4.8) | 3.8 (2.7)

10. Secondary Outcome: Worst Leg Pain Score
Description: Worst leg pain score on 0-10 numerical rating scale over the last week (higher pain scores indicate greater pain)
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 4.9 (3.3) | 4.8 (3.4) | 5.8 (2.9)

11. Secondary Outcome: Average Back Pain Score
Description: Average back pain score on 0-10 numerical rating scale over the last week (higher pain scores indicate greater pain)
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 3.1 (2.3) | 3.5 (2.6) | 3.6 (2.7)

12. Secondary Outcome: Worst Back Pain Score
Description: Worst back pain score on 0-10 numerical rating scale over the last week (higher pain scores indicate greater pain)
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 5.1 (3.5) | 5.5 (3.3) | 5.5 (3.1)

13. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Patient global impression of change on 7-point Likert scale (from 1= no change, 3= a little better 5= moderately better, a slight but noticeable change, to 7=a great deal better, a considerable improvement that has made all the difference)
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 4.7 (1.8) | 4.5 (2.0) | 4.6 (1.9)

14. Secondary Outcome: Number of Participants With Analgesic Reduction
Description: Categorical reduction in analgesic usage (cessation of non-opioid analgesic and/ or > 20% reduction in opioid use)
Time Frame: 4 weeks
Population: Five participants were lost to follow-up and did not have 4 weeks outcomes measured. Eleven participants did not have data recorded for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 46 | 44 | 40
Participants | 16 | 19 | 7

15. Secondary Outcome: Oswestry Disability Index (ODI) Score
Description: Functional measurement of back and leg pain disability on 0-100% scale (higher levels indicate greater disability)
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 32 (17) | 36 (17) | 34 (15)

16. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Scores for Anxiety and Depressions
Description: The Hospital anxiety and depression scale (HADS) is an instrument used to measure depression and anxiety. Anxiety and depression are scored separately, each on a subscale. The score on each subscale ranges from 0 to 21 score on a scale. A score of 0 indicates the absence of depression or anxiety. A score of 21 indicated severe depression or anxiety. The subscales are not combined for a total score. Anxiety score is reported.
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 4.9 (4.0) | 5.1 (4.5) | 4.3 (3.0)

17. Secondary Outcome: Number of Participants With Complications
Description: Number of Participants With Complications related to the procedure, sedation or use of virtual reality
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 50 | 48
Participants | 5 | 10 | 4

18. Secondary Outcome: Percentage Change of the Spectral Edge Frequency (SEF)
Description: Frontal EEG sensor will be placed with electrode positions corresponding to Fp1, Fp2, F7, and F8 in the international 10-20 system. The spectral edge frequency (SEF) on the Sedline monitor ranges in frequency from 0 to 30 Hz.
Time Frame: During the procedure for up to 20 minutes
Population: The bifrontal EEG was used in an arbitrary subgroup of participants based on the availability of the EEG.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 4 | 6 | 6
percentage change | 0.56 (5.44) | 64.05 (44.35) | 53.43 (19.16)

19. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Scores for Depression and Anxiety
Description: The Hospital anxiety and depression scale (HADS) is an instrument used to measure depression and anxiety. Anxiety and depression are scored separately, each on a subscale. The score on each subscale ranges from 0 to 21 score on a scale. A score of 0 indicates the absence of depression or anxiety. A score of 21 indicated severe depression or anxiety. The subscales are not combined for a total score. Depression score is reported.
Time Frame: 4 weeks
Population: Participants who completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
Number analyzed (Participants) | 48 | 48 | 45
score on a scale | 4.0 (3.9) | 4.5 (3.9) | 3.8 (3.5)

ADVERSE EVENTS:
Time Frame: Up to 4 weeks post-procedure
Arm/Group | Virtual Reality (VR) | Sedation | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 5/48 | 10/50 | 4/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Virtual Reality (VR) (N=48) | Sedation (N=50) | Standard Care (N=48)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) — Nausea
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Vomiting
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) — Respiratory Depression
Dizziness (Ear and labyrinth disorders) | 1 (1) | 3/3 (3) | 1 (1) — Dizziness
Severe pain (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) — Severe pain
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — Tachycardia
Diaphoresis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Diaphoresis
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Shingles
Procedure site swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Procedure site swelling
Dural Puncture (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Dural Puncture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04887285/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT04887285/ICF_001.pdf